CLINICAL TRIAL: NCT05021900
Title: A Phase II, Multi-center, Randomized, Open-label, Two-arm Study to Assess the Efficacy and Safety of Tenalisib (RP6530), a PI3K δ/γ and SIK3 Inhibitor, in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Efficacy and Safety of Tenalisib (RP6530), in Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-2101
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: RP6530; Tenalisib
MeSH Terms: conditions — Breast Neoplasms | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenalisib 800 mg BID (Experimental): Single agent at a dose of 800 mg BID
  Interventions: Drug: Tenalisib 800mg
- Tenalisib 1200 mg BID (Experimental): Single agent at a dose of 1200 mg BID
  Interventions: Drug: Tenalisib 1200mg

INTERVENTIONS:
Drug: Tenalisib 800mg — Tenalisib will be administered 800mg BID, orally
  Other Names: RP6530
  Arms: Tenalisib 800 mg BID
Drug: Tenalisib 1200mg — Tenalisib will be administered 1200mg BID, orally
  Other Names: RP6530
  Arms: Tenalisib 1200 mg BID

SUMMARY:
Phase II, randomized, open-label study, designed to evaluate the preliminary efficacy and safety of tenalisib at two dose levels in 40 patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
The study will have two groups, Group 1 with a treatment option of 800mg RP6530 BID and Group 2 with a treatment option of 1200mg RP6530 BID, where the subjects will be randomly assigned to each group in 1:1 and continued on each group of treatment till disease progressed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years of age, at the time of signing informed consent.
2. Female patients who have histologically and/or cytologically confirmed locally advanced or metastatic breast cancer that has progressed following at least one line of therapy.
3. Patients with at least one measurable lesion per RECIST version 1.1 at baseline that can be accurately assessed by CT scan or MRI and is suitable for repeated assessment at follow up-visits.
4. ECOG performance status 0 to 2.
5. Life expectancy of at least 3 months.
6. Adequate bone marrow, liver, and renal functions
7. Female patients of childbearing potential should be willing to use a medically acceptable method of contraception

Exclusion Criteria:

1. Patients with HER-2 positive breast cancer.
2. Patients receiving anticancer therapy within 4 weeks or 5 half-lives of the drug prior to C1D1, whichever is shorter.
3. Patient who has not recovered from acute toxicities (defined as NCI-CTCAE grade > 1) of previous therapy except treatment-related alopecia.
4. Patients who have had disease progression within 8 weeks of platinum chemotherapy.
5. Prior exposure to investigational or marketed PI3K inhibitors given for the treatment of breast cancer.
6. Major surgery within 4 weeks of starting study treatment OR any patient who has not recovered from the effects of major surgery.
7. Patient with symptomatic uncontrolled brain metastasis.
8. HIV-positive patients who are on antiretroviral therapy OR active hepatitis C OR active hepatitis B virus infections.
9. Ongoing immunosuppressive therapy including systemic corticosteroids except as allowed per concomitant medication.
10. Known history of severe liver injury as judged by the investigator.
11. History of severe cutaneous reactions in the past.
12. Active gastrointestinal tract disease with malabsorption syndrome or uncontrolled inflammatory gastrointestinal disease such as Crohn's disease or ulcerative colitis.
13. Pregnancy or lactation.
14. Patient with other active malignancies at the time of screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (3):
  - High Technology Hospital Medcenter, Batumi
  - LLC Caucasus Medical Center, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenalisib 800 mg BID: Tenalisib: Tenalisib will be administered 800mg BID, orally
- Tenalisib 1200 mg BID: Tenalisib: Tenalisib will be administered 1200mg BID, orally
Period: Overall Study
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 61.27 [31.10 to 71.47] | 64.21 [51.95 to 71.71] | 63.18 [31.10 to 71.71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Georgia | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Without Disease Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Approximately 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Tenalisib 800 mg BID: Tenalisib was be administered 800mg BID, orally
- Tenalisib 1200 mg BID: Tenalisib was administered 1200mg BID, orally
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Number analyzed (Participants) | 20 | 20
Participants | 7 | 8

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Approximately 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Number analyzed (Participants) | 20 | 20
Participants | 2 | 3

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: It is defined as sum of CR, PR and SD rates
Time Frame: Approximately 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Number analyzed (Participants) | 20 | 20
Participants | 11 | 12

4. Secondary Outcome: Progression Free Survival (PFS).
Description: PFS is measured from the time of first dose of study drug to radiographic documentation of disease progression or death due to any cause.
Time Frame: Approximately 18 months
Measure: Median (Full Range); unit: days
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Number analyzed (Participants) | 16 | 19
days | 170 [29 to 513] | 170 [38 to 454]

5. Secondary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product.
Time Frame: Approximately 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
Number analyzed (Participants) | 20 | 20
Participants | 15 | 17

ADVERSE EVENTS:
Time Frame: Approximately 18 months
Arm/Group | Tenalisib 800 mg BID | Tenalisib 1200 mg BID
All-Cause Mortality (participants affected / at risk) | 2/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 5/20 | 1/20
Other Adverse Events (participants affected / at risk) | 15/20 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib 800 mg BID (N=20) | Tenalisib 1200 mg BID (N=20)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib 800 mg BID (N=20) | Tenalisib 1200 mg BID (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1 (5) | 3 (6)
Fatigue (General disorders) | 1 (1) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 8 (21) | 12 (20)
Alanine aminotransferase increased (Investigations) | 8 (16) | 10 (13)
Aspartate aminotransferase increased (Investigations) | 8 (14) | 8 (12)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (8) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This is an open label study in a limited number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT05021900/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05021900/SAP_001.pdf